CLINICAL TRIAL: NCT00195416
Title: A Drug Use Investigation of Enbrel for Post-marketing Surveillance (PMS) for Ankylosing Spondylitis
Brief Title: Study Investigating Enbrel Treatment for Ankylosing Spondylitis
Status: Completed | Type: Observational
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Other Study IDs: 0881A-102018
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2009-09-16 (Estimated); Status verified 2009-09

CONDITIONS: Ankylosing Spondylitis
Keywords: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Etanercept

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Etanercept — Etanercept 25mg Injection, 2 times/week

SUMMARY:
To identify the following problems and questions with respect to the safety and effectiveness of Enbrel during the post-marketing period as required by Korea Food and Drug Administration (KFDA)'s regulations.

1. Unknown adverse reactions, especially serious adverse reactions
2. Change of the incidences of adverse reactions under the routine drug uses
3. Factors that may affect the safety of the drug
4. Factors that may affect the effectiveness of the drug

ELIGIBILITY:
Inclusion Criteria:

* Adults: Severe ankylosing spondylitis (AS) in patients who do not respond adequately to previous therapy

Exclusion Criteria:

* Patients with known hypersensitivity to Enbrel or any component of the product
* Patients with sepsis or risk of sepsis
* Patients with active infections including chronic or localized infections such as tuberculosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic, secondary and tertiary medical centers
Sampling Method: Non-Probability Sample
Enrollment: 526 (Actual)
Dates: Start 2005-06; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (2):
- South Korea (2):
  - Gyunggi-do
  - Seoul